CLINICAL TRIAL: NCT01976663
Title: A Prospective, Multicenter, Within-subject Controlled Study of the Safety and Effectiveness of JUVÉDERM VOLIFT® XC Versus Control for the Correction of Moderate to Severe Nasolabial Folds
Brief Title: A Safety and Effectiveness Study of JUVÉDERM VOLIFT® XC Versus Control for Moderate to Severe Nasolabial Folds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allergan (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: S17L-001
Record Dates: First submitted 2013-10-30; First posted 2013-11-06 (Estimated); Results first posted 2017-05-22 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-03

CONDITIONS: Moderate to Severe Nasolabial Folds

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- VOLIFT® XC NLFs (Experimental): Nasolabial folds treated with JUVEDERM VOLIFT® XC.
  Interventions: Device: JUVEDERM VOLIFT® XC
- Control NLFs (Active Comparator): Nasolabial folds treated with Control.
  Interventions: Device: Control

INTERVENTIONS:
Device: JUVEDERM VOLIFT® XC — Up to 4 mLs JUVEDERM VOLIFT® XC injected intradermally in one NLF (total; including initial and touch-up treatments) and up to 4 mLs JUVEDERM VOLIFT XC is allowed for repeat treatment. For asymmetric correction, only the more severe NLF is eligible for asymmetric correction.
  Arms: VOLIFT® XC NLFs
Device: Control — Up to 4 mLs Control injected intradermally in opposite NLF (total; including initial and touch-up treatments). Up to 4 mLs JUVEDERM VOLIFT XC is allowed for asymmetry correction and up to 4 mLs JUVEDERM VOLIFT XC is allowed for repeat treatment. Only the more severe NLF is eligible for asymmetric correction.
  Arms: Control NLFs

SUMMARY:
A prospective, multicenter, within-subject controlled study of the safety and effectiveness of JUVÉDERM VOLIFT® XC versus Control for the correction of moderate to severe nasolabial folds (NLFs).

ELIGIBILITY:
Inclusion Criteria:

* 2 visible moderate to severe nasolabial folds
* Agree to refrain from undergoing other anti-wrinkle/volumizing treatments in the lower two-thirds of the face for the duration of the study

Exclusion Criteria:

* Undergone facial tissue augmentation with dermal fillers in the lower two-thirds of the face within the past 12 months
* Undergone facial tissue augmentation with fat injections, botulinum toxin injections in the lower two-thirds of the face, mesotherapy, or cosmetic facial procedures in the face or neck within the past 6 months
* Received semi-permanent fillers or permanent facial implants anywhere in the lower face

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2013-10-29 (Actual); Primary Completion 2015-03-17 (Actual); Study Completion 2015-10-26 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Total Skin and Beauty Dermatology Center P.C., Birmingham, Alabama
  - Vitiligo and Pigmentation Institute of Southern California, Los Angeles, California
  - San Francisco, California
  - Dermatology Research Institute, LLC, Coral Gables, Florida
  - Skin Research Institute, Coral Gables, Florida
  - West Palm Beach, Florida
  - Chicago, Illinois

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Monheit G, Beer K, Hardas B, Grimes PE, Weichman BM, Lin V, Murphy DK. Safety and Effectiveness of the Hyaluronic Acid Dermal Filler VYC-17.5L for Nasolabial Folds: Results of a Randomized, Controlled Study. Dermatol Surg. 2018 May;44(5):670-678. doi: 10.1097/DSS.0000000000001529. PMID 29701621

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 126 subjects were enrolled (Enrolled Population); 123 subjects were randomized and treated (Modified Intent-to-Treat). Each subject had one nasolabial fold treated with JUVEDERM VOLIFT® XC and one treated with control. After initial treatment, subjects were eligible for touch-up, asymmetry correction, and repeat treatment per protocol.
Groups:
- JUVEDERM VOLIFT® XC: Nasolabial folds treated with JUVEDERM VOLIFT® XC on one side and Control on the other side.
Period: Overall Study
Arm/Group | JUVEDERM VOLIFT® XC
Started | 126
Received Touch-up Treatment | 63
Received Asymmetry Correction | 45
Received Repeat Treatment | 85
Completed | 84
Not Completed | 42
Not completed — Completed 18 mos but no repeat treatment | 24
Not completed — Personal Reasons | 6
Not completed — Withdrawal by Subject | 4
Not completed — Screen Failure | 3
Not completed — Adverse Event | 2
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Modified Intent-to-Treat (mITT): all randomized and treated subjects
Arm/Group | JUVEDERM VOLIFT® XC
Number analyzed (Participants) | 123
Age, Customized [Count of Participants; unit: Participants]
  30 to 50 years | 36
  51 to 65 years | 72
  >65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 117
  Male | 6

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Nasolabial Fold Severity Using the 5-Point Nasolabial Fold Severity Scale (NLFSS)
Description: Nasolabial fold severity is assessed by the Evaluating Investigator on the 5-point Nasolabial Fold Severity Scale (ranging from 0=None [no wrinkle] to 4=Extreme [very deep wrinkle, redundant fold]). Mean change from baseline in NFLSS is defined as score at baseline minus score at Month 6. A negative number change from baseline indicated improvement and a positive number change from baseline indicated worsening.
Time Frame: Baseline, Month 6
Population: modified intent-to-treat (mITT): all randomized and treated subjects
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Groups:
- JUVEDERM VOLIFT® XC: Nasolabial folds treated with JUVEDERM VOLIFT® XC.
- Control: Nasolabial folds treated with Control.
Arm/Group | JUVEDERM VOLIFT® XC | Control
Number analyzed (Participants) | 123 | 123
Scores on a Scale
  Baseline | 2.6 (0.49) | 2.6 (0.49)
  Month 6 (N=117, 117): number analyzed (Participants) | 117 | 117
  Month 6 (N=117, 117) | 1.4 (0.67) | 1.3 (0.72)

2. Primary Outcome: Percentage of Nasolabial Folds With ≥1-Point Improvement
Description: Nasolabial fold severity is evaluated by the Evaluating Investigator on the 5-point Nasolabial Fold Severity Scale (ranging from 0=None [no wrinkle] to 4=Extreme [very deep wrinkle, redundant fold]). The percentage of nasolabial folds with ≥1-point improvement from baseline (i.e., decrease in severity) are reported.
Time Frame: Baseline, Month 6
Population: modified intent-to-treat (mITT): all randomized and treated subjects with data for this outcome measure
Measure: Number (95% Confidence Interval); unit: Percentage of Nasolabial Folds
Arm/Group | JUVEDERM VOLIFT® XC | Control
Number analyzed (Participants) | 117 | 117
Percentage of Nasolabial Folds | 93.2 (0.49) [87.0 to 97.0] | 86.3 [78.7 to 92.0]

3. Secondary Outcome: Percentage of Nasolabial Folds With ≥1-Point Improvement
Description: as for outcome 2
Time Frame: Baseline, Month 12
Population: modified intent-to-treat (mITT): all randomized and treated subjects with data for this outcome measure
Measure: Number (95% Confidence Interval); unit: Percentage of Nasolabial Folds
Arm/Group | JUVEDERM VOLIFT® XC | Control
Number analyzed (Participants) | 113 | 113
Percentage of Nasolabial Folds | 57.5 (0.49) [47.9 to 66.8] | 56.6 [47.0 to 65.9]

4. Secondary Outcome: Mean Change From Baseline in Overall Nasolabial Folds FACE-Q Score
Description: Subjects evaluate nasolabial folds on the 5-item Nasolabial Folds module of the FACE-Q questionnaire. Responses to the 5 items are combined to create a scale score that ranged from 0 to 100, where 0 indicates that the subject is extremely bothered and 100 indicates that the subject is not all bothered by the appearance of the nasolabial fold. Change from baseline is defined as the score at Month 12 minus the baseline score. A positive number change from baseline indicates an improvement and a negative number change from baseline indicates a worsening.
Time Frame: Baseline, Month 12
Population: modified intent-to-treat (mITT): all randomized and treated subjects with data at this time point
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | JUVEDERM VOLIFT® XC | Control
Number analyzed (Participants) | 123 | 123
Scores on a Scale
  Baseline | 32.1 (14.70) | 32.0 (14.94)
  Month 12 (N=112, 111): number analyzed (Participants) | 112 | 111
  Month 12 (N=112, 111) | 25.8 (23.08) | 23.4 (22.83)

ADVERSE EVENTS:
Description: The Safety Population includes all subjects who received at least 1 treatment. The Safety Population is used to assess adverse events and serious adverse events. Adverse events and serious adverse events are presented by treatment side for events occurring at the nasolabial folds, or combined for events that did not occur at the nasolabial folds.
Groups:
- JUVEDERM VOLIFT® XC During Initial/Touch Up: Nasolabial folds treated with JUVEDERM VOLIFT® XC during the Initial/Touch Up period.
- Control During Initial/Touch Up Treatment Period: Nasolabial folds treated with Control during the Initial/Touch Up period.
- Not at NLF During Initial/Touch Up Treatment Period: Nasolabial folds treated with JUVEDERM VOLIFT® XC on one side and Control on the other side.
- JUVEDERM VOLIFT® XC Asymmetry Correction/Repeat Treatment: Nasolabial folds treated with JUVEDERM VOLIFT® XC during the Asymmetry Correction/Repeat Treatment period.
Arm/Group | JUVEDERM VOLIFT® XC During Initial/Touch Up | Control During Initial/Touch Up Treatment Period | Not at NLF During Initial/Touch Up Treatment Period | JUVEDERM VOLIFT® XC Asymmetry Correction/Repeat Treatment
Serious Adverse Events (participants affected / at risk) | 0/123 | 0/123 | 5/123 | 0/93
Other Adverse Events (participants affected / at risk) | 29/123 | 27/123 | 0/123 | 19/93
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | JUVEDERM VOLIFT® XC During Initial/Touch Up (N=123) | Control During Initial/Touch Up Treatment Period (N=123) | Not at NLF During Initial/Touch Up Treatment Period (N=123) | JUVEDERM VOLIFT® XC Asymmetry Correction/Repeat Treatment (N=93)
Cardiac Arrest (Cardiac disorders) | 0 | 0 | 1 | 0 — Subject 10003-3015; occurred 1 year after treatment; assessed as unrelated to treatment
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0 — Assessed as unrelated to treatment
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 0 — Subject 10003-3015; occurred 1 year after treatment; assessed as unrelated to treatment
Basal Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 — Assessed as unrelated to treatment
Squamous Cell Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 — Assessed as unrelated to treatment
Brain Hypoxia (Nervous system disorders) | 0 | 0 | 1 | 0 — Subject 10003-3015; occurred 1 year after treatment; assessed as unrelated to treatment
Cerebrovascular Accident (Nervous system disorders) | 0 | 0 | 1 | 0 — Subject 10003-3015; occurred 1 year after treatment; assessed as unrelated to treatment
Seizure (Nervous system disorders) | 0 | 0 | 1 | 0 — Subject 10003-3015; occurred 1 year after treatment; assessed as unrelated to treatment
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 — Subject 10003-3015; occurred 1 year after treatment; assessed as unrelated to treatment
Ovarian Cyst (Reproductive system and breast disorders) | 0 | 0 | 1 | 0 — Assessed as unrelated to treatment
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | JUVEDERM VOLIFT® XC During Initial/Touch Up (N=123) | Control During Initial/Touch Up Treatment Period (N=123) | Not at NLF During Initial/Touch Up Treatment Period (N=123) | JUVEDERM VOLIFT® XC Asymmetry Correction/Repeat Treatment (N=93)
Injection Site Induration (General disorders) | 13 | 11 | 0 | 10
Injection Site Mass (General disorders) | 9 | 9 | 0 | 9
Injection Site Swelling (General disorders) | 9 | 9 | 0 | 3
Injection Site Bruising (General disorders) | 5 | 1 | 0 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
A disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 90 days from the time submitted to the sponsor for review. The sponsor cannot require changes to the communication and cannot extend the embargo.